CLINICAL TRIAL: NCT02285218
Title: Role of New Adipokines and Hepatokines in Prediction of Patients With Metabolic Syndrome or NAFLD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2014-0073
Record Dates: First submitted 2014-11-04; First posted 2014-11-06 (Estimated); Last update posted 2019-03-18 (Actual); Status verified 2019-03

CONDITIONS: Non-alcoholic Fatty Liver Disease; Type 2 Diabetes; Metabolic Syndrome
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Diabetes Mellitus, Type 2; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma (blood)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- 1) Normal control: metabolically healthy with no obesity
  Interventions: Other: serum blood sampling
- 2) dyslipidemia: high triglyceride levels or LDL-C levels
  Interventions: Other: serum blood sampling
- 3) type 2 diabetes: defined in 'inclusion criteria'
  Interventions: Other: serum blood sampling
- 4) non-alcoholic fatty liver disease: defined in 'inclusion criteria'
  Interventions: Other: serum blood sampling

INTERVENTIONS:
Other: serum blood sampling

SUMMARY:
To investigate the predictive roles of adipokines and hepatokines to detect non-alcoholic fatty liver disease (NAFLD), diabetes, or dyslipidmia.

To examine the association or effects of clinical and biochemical factors (lab results and medication, etc.) on serum levels of adipokines and hepatokines in certain subjects with non-alcoholic fatty liver disease (NAFLD), diabetes, or dyslipidmia.

ELIGIBILITY:
Inclusion Criteria:

1. dyslipidemia 1. serum triglyceride≥150mg/dl, or taking medication to lower triglyceride levels (e.g. fibrates, niacin, omega-3, etc.) or 2. serum LDL-C≥100mg/dl, or taking medication to lower LDL-C levels (e.g. statin, ezetimibe, etc.)
2. type 2 diabetes 1. defined according to the ADA guideline (DM definition) or 2. taking any anti-diabetic medications
3. non-alcoholic fatty liver disease (NAFLD) 1. diagnosed as having fatty liver by ultrasonogram or 2. diagnosed as having fatty liver by transient elastogram (Fibroscan) or 3. diagnosed as having fatty liver by abdomina CT scan
4. Normal control 1. should not be included in other groups as above and 2. not taking any medication related to diabetes and dyslipidemia and 3. BMI <25kg/m2

Exclusion Criteria:

1. subjects who refused to agree with informed consents
2. subjects with organ-transplantation
3. serum creatinine ≥1.5mg/dl
4. pregnant women
5. liver cancer or pancreatic cancer
6. subjects with chronic hepatitis B or C virus infection
7. for NAFLD group, subjects with excessive alcohol consumption (men: ≥210g of alcohol per week, women: ≥140g of alcohol per week)

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects are recruited from either patients who visit out-patient clinics (Diabetes center in Severance hospital) or healthy volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2014-04; Primary Completion 2019-03 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
new adipokines | To 8h fasting blood sample
  several candidate adipokines and hepatokines to predict diseases will be measured using ELISA
new hepatokines | To 8h fasting blood sample
  several candidate adipokines and hepatokines to predict diseases will be measured using ELISA

CONTACTS AND LOCATIONS:
Locations (1):
- Severance hospital, Seoul, South Korea

REFERENCES:
- [Derived] Lee YH, Lee SG, Lee CJ, Kim SH, Song YM, Yoon MR, Jeon BH, Lee JH, Lee BW, Kang ES, Lee HC, Cha BS. Association between betatrophin/ANGPTL8 and non-alcoholic fatty liver disease: animal and human studies. Sci Rep. 2016 Apr 5;6:24013. doi: 10.1038/srep24013. PMID 27045862